CLINICAL TRIAL: NCT05009615
Title: Efficacy of New Products Combining Hydroxycinnamates and Beta-glucans as a Dietary Tool Against Obesity and Associated Dysfunctions (Hyperglycemia and Dyslipemia)
Brief Title: Efficacy of Hydroxycinnamates and Beta-glucans as a Dietary Tool Against Obesity (OBHEALTH)
Acronym: OBHEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Laura Bravo, Professor, Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AGL2015-69986-R
Record Dates: First submitted 2021-07-29; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Overweight/Obesity; Insulin Resistance
Keywords: Obesity; Non-communicable diseases; Polyphenols; Soluble dietary fiber; Nutraceutical
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Noncommunicable Diseases | interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: After a run-in period, participants were randomly allocated to one of each arm. Each intervention stage (8 weeks) was separated by a 4-week wash-out.
Who Masked: Participant
Masking Description: Nutraceutical was provided in aluminum foil sachets marked A, B or C for blinding to participants. Aroma and flavor compounds were added to ensure similar organoleptic properties of the 3 nutraceuticals tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Green coffee extract (Experimental): Nutraceutical containing a decaffeinated green coffee extract rich in phenolic compounds (hydroxycinnamates). Participants received powdered sachets containing 300 mg of GC extract twice daily for 8 weeks
  Interventions: Dietary Supplement: Green coffee extract
- Beta-glucan (Experimental): Nutraceutical containing a oat beta-glucan. Participants received powdered sachets containing 2.5 g of BG twice daily for 8 weeks
  Interventions: Dietary Supplement: Beta glucan
- Green coffee + Beta-glucan (Experimental): Nutraceutical containing both green coffee extract and beta-glucan. Participants received powdered sachets containing 2.5 g of BG plus 300 mg of GC extract twice daily for 8 weeks
  Interventions: Dietary Supplement: Green coffee + beta-glucan

INTERVENTIONS:
Dietary Supplement: Green coffee extract — 150 mg polyphenols from green coffee, twice daily
  Arms: Green coffee extract
Dietary Supplement: Beta glucan — 2.5 g BG twice daily
  Arms: Beta-glucan
Dietary Supplement: Green coffee + beta-glucan — 150 mg polyphenols from green coffee + 2.5 g BG, twice daily
  Arms: Green coffee + Beta-glucan

SUMMARY:
The study aimed at assessing the effect of a decaffeinated green coffee extract, rich in hydroxycinnamates, oat beta-glucans or the combination of both bioactive compounds on overweight/obese subjects with hyperglycemia.

DETAILED DESCRIPTION:
In a randomized, crossover, blind, three-arm study, volunteers consumed twice a day a nutraceutical providing 5 g/d beta-glucan (BG), 600 mg/d green coffee polyphenols (GC) or a combination of both (5 g/d BG + 600 mg/d GC). Each intervention stage lasted 8 weeks and was followed by a 4-week wash-out.

Blood, urine and fecal samples were obtained at the beginning and end of each intervention stage. Blood pressure, oral glucose tolerance test (OGTT) and body composition (body weight, anthropometry, bioimpedance) were measured at each control visit. Physical activity was controlled by accelerometry (1 week during each intervention stage). Energy expenditure was measured by calorimetry. Food intake was monitored by 3-d food records. Satiety was determined by subjective (VAS) and objective (weighting consumed food) records after consuming the nutraceutical during each intervention stage.

In a subset of volunteers (9), a pharmacokinetic study was performed to assess bioavailability and metabolism of polyphenols at the beginning and end of each intervention (GC and GC+BG only). In these volunteers, blood was taken at different times during 24 h; urine samples were also collected at different intervals during 24 h, and feces were obtained at 0 and 24 h approximately after consuming the nutraceuticals containing GC. A targeted metabolomic analysis was carried out in these samples. In these volunteers, incretins and hormones were also determined in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, with BMI between 25-35 kg/m2
* Fasting blood glucose between 6,11-6,94 mmol/L (110-125 mg/dL) and/or
* Blood glucose between 7,77-11,04 mmol/L (140-199 mg/dL) 2 h after an oral glucose overload

Exclusion Criteria:

* Having other chronic pathologies different from overweight/obesity and prediabetes.
* On prescription drugs, hormones or dietary supplements (e.g. dietary fibre, pollen, vitamin complexes, etc.)
* Vegetarian
* Smoking
* Known hypersensibility/allergy to any of the tests products
* Pregnant women
* On dietary regimen or physical training to lose weight

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Body weight | 8 weeks
  Change of body weight (estimated 2.5 kg) at the end of the intervention

SECONDARY OUTCOMES:
Body fat percentage | 8 weeks
  Change of body fat percentage (total and visceral)
Anthropometry | 8 weeks
  Change of body circumferences (waist, hip, thigh) or skin folds at the end of the intervention
Insulin resistance | 8 weeks
  Change in fasting blood glucose and/or insulin levels, use to calculate homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR), beta-cell function (HOMA-beta) or quantitative insulin sensitivity check index (QUICKI) indexes. Outcome would be a modification of at least one of these indexes at the end of the intervention
Blood lipids | 8 weeks
  Modification of serum levels of total cholesterol, LDL-cholesterol, HDL-cholesterol blood, triglycerides at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bravo, Prof, Principal Investigator — ICTAN-CSIC
Locations (1):
- Instituto de Ciencia y Tecnología de Alimentos y Nutrición, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No